CLINICAL TRIAL: NCT01592838
Title: Feasibility Pilot Study Assessing the Impact on the Quality of Hospital Care After the Introduction of Rotavirus Vaccination in Belgium
Brief Title: Impact on Quality of Hospital Care During Pre- and Post- Rotavirus (RV) Vaccination Introduction in Belgium
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 116721
Record Dates: First submitted 2012-05-03; First posted 2012-05-07 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Infections, Rotavirus
Keywords: Belgium; Quality of hospital care; Rotavirus vaccination
MeSH Terms: conditions — Rotavirus Infections | interventions — Data Collection

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Hospitalized Group: Data collection for changes in hospital pattern pre- versus post-rotavirus vaccination, in children ≤15 years old hospitalised for any reason between June 2004 and May 2010.
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — The participating centre will be requested to generate a coded list of all hospitalisations taken place during the study period (June 1st 2004- May 31st 2010) and analysed for changes in hospital pattern pre- versus post-rotavirus vaccination, in children aged ≤15 years.

SUMMARY:
This study aims to investigate whether a change in the pattern of hospitalisation was observed in paediatric wards over the last 6 years (June 2004 - May 2010), whether a change in staff workforce availability was observed in paediatric wards over the last 6 years (during a whole year or during specific time periods of the year) and if changes of any of the variables measured during the observation period could be linked to the introduction of rotavirus vaccination.

DETAILED DESCRIPTION:
This retrospective study will use data extracted from hospital databases during the period of the 1st of June 2004 until the 31st of May 2010. A coded list of all hospitalisations and of the different infection tests performed in children will be generated, together with a list of Full time equivalents (FTE) in paediatric ward and the number of sick leave days of the working personnel.

ELIGIBILITY:
Inclusion Criteria:

* All children aged ≤15 years being hospitalised (with overnight stay or day clinic) for whatever reason during the study period

Exclusion Criteria:

* Not Applicable

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children ≤15 years old hospitalised for any reason between June 2004 and May 2010.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2013-12; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Determination of changes in hospitalisation pattern and workforce availability at the level of a pediatric ward in a hospital setting. | During the study period (from June 1st 2004 up to 6 years)

SECONDARY OUTCOMES:
Expression of the changes into a quality of hospital care score that can be easily applied in different hospital settings. | During the study period (from June 1st 2004 up to 6 years)
Determination through factor and regression analysis which variable influences most the score in order to improve the score calculation. | During the study period (from June 1st 2004 up to 6 years)
Investigation of whether a change in the quality of hospital care score could be linked to the introduction of rotavirus vaccination. | During the study period (from June 1st 2004 up to 6 years)
Observation of other changes in the hospital organisation as a consequence of a change in the quality of hospital care score. | During the study period (from June 1st 2004 up to 6 years)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline